CLINICAL TRIAL: NCT00592774
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Tolerability Titration Study To Evaluate The Efficacy And Safety Of Perampanel (E2007) In Patients With Post-Herpetic Neuralgia (PHN)
Brief Title: Dose-Tolerability Titration Study to Evaluate The Efficacy And Safety Of Perampanel (E2007) In Patients With Post-Herpetic Neuralgia (PHN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2007-A001-218
Record Dates: First submitted 2008-01-03; First posted 2008-01-14 (Estimated); Results first posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Neuralgia
Keywords: Post-Herpetic Neuralgia; PHN)
MeSH Terms: conditions — Neuralgia; Neuralgia, Postherpetic | interventions — perampanel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Placebo Cohort 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- Perampanel Cohort 1, 3-week Titration (Experimental)
  Interventions: Drug: E2007 (perampanel)
- Placebo Cohort 2 (Experimental)
  Interventions: Drug: Placebo
- Perampanel Cohort 2, 1-week Titration (Experimental)
  Interventions: Drug: E2007 (perampanel)
- Perampanel Cohort 2, 2- Week Titration (Experimental)
  Interventions: Drug: E2007 (perampanel)

INTERVENTIONS:
Drug: E2007 (perampanel) — 2 mg titrated up to 8 mg maximum; taken once daily.
  Other Names: perampanel
  Arms: Perampanel Cohort 1, 3-week Titration; Perampanel Cohort 2, 1-week Titration; Perampanel Cohort 2, 2- Week Titration
Drug: Placebo — 2 mg titrated up to 8 mg maximum; taken once daily.
  Arms: Placebo Cohort 1; Placebo Cohort 2

SUMMARY:
The purpose of the study is to determine the efficacy and safety of Perampanel (E2007) in patients with Post-Herpetic Neuralgia (PHN).

ELIGIBILITY:
Inclusion Criteria:

To be included, patients must meet the following:

1. Provide written informed consent, prior to entering the study or undergoing any study procedures.
2. Male and female patients ≥18 years of age. Females should be either of nonchildbearing potential as a result of surgery or menopause (1 year after onset), or of childbearing potential and practicing a medically acceptable method of contraception. Acceptable contraception includes: abstinence, a barrier method plus spermicide, or intrauterine device [IUD]. Those females using hormonal contraceptives must also be using an additional approved method of contraception (e.g., a barrier method plus spermicide or IUD). Contraceptive use must start at least 1 month before Visit 1, be practiced throughout the entire study period, and continue for 1 month after the end of the study. They must also have a negative serum beta-human chorionic gonadotropin (β-hCG) at Visit 1, and a negative urine pregnancy test at Baseline Visit 2.
3. PHN of at least 6 months duration; the onset of PHN is defined as the time from healing of herpes zoster skin lesions.
4. Pain over the past 6 months, and not in a clinically identifiable improving or worsening trend, based on medical history.
5. Score of ≥ 40 mm on the visual analog scale (VAS) of the short form McGill Pain Questionnaire (SF-MPQ) at both Visit 1 and Baseline (Visit 2 prior to randomization).
6. Have completed the patient diary for at least 6 of the 7 days prior to Visit 2 (Baseline).
7. Average daily pain score of ≥ 4, on 11-point Likert scale during the 7 days prior to randomization [from the diaries].
8. Reliable and willing and able to cooperate with all study procedures, including the following examples:

   * Accurately entering the diary on a daily basis
   * Returning for study visits on the required dates
   * Accurately and reliably reporting symptoms (including treatment-emergent signs and symptoms)
   * Taking study drug as required by protocol
9. Be on stable analgesic treatment (same medication(s)) or stable nonpharmacological pain treatment for at least 4 weeks prior to Visit 1 and remain on this stable treatment throughout the study. Nonpharmacologic pain treatment includes the following:

   * relaxation/hypnosis
   * physical or occupational therapy
   * mental-health counseling
   * acupuncture
   * injections
   * blocks, etc.
   * Episodic or periodic pharmacologic treatments such as monthly injections for treatment of pain (eg, local anesthetics) will not be permitted.
   * Up to 4 g of acetaminophen/day is permitted as rescue medication, as needed, during the trial.

Exclusion Criteria:

Patients with any of the following are to be excluded:

1. Any condition that could interfere with the conduct of the trial or confound efficacy evaluations including the following examples: pain or neuropathy from another cause (including painful diabetic neuropathy), such as central pain, radiculopathy, painful arthritis, etc.
2. Motivation by secondary gain, or where there is a negative-incentive to achieving pain and functional relief (eg, litigation). This will be determined from the medical history and is at the discretion of the investigator.
3. Inability to cooperate with protocol, for any reason.
4. Clinically significant, progressive, or potentially unstable disease of any body system including cardiovascular, gastrointestinal, CNS, psychiatric, endocrine, or immunologic, including patients with any of the following broad disease categories:

   1. Systemic infections (eg, human immunodeficiency virus [HIV], hepatitis, tuberculosis [TB], syphilis); lack of appropriate medical history of these conditions is acceptable,
   2. History of past (within the past 12 months) or present drug or alcohol abuse as per the Diagnostic and Statistical Manual - 4th Edition (DSM IV) criteria,
   3. History of acute coronary syndrome within the past 12 months,
   4. Active cancer within the previous 5 years (the exception is fully treated, non-melanoma skin cancer such as basal cell carcinoma),
   5. Systemic chemotherapy or immunotherapy within the past 5 years,
   6. History of major depression, bipolar disease, psychosis or suicidal ideation or attempts within the past 5 years,
   7. History of major systemic allergy such as anaphylactoid reactions or Stevens-Johnson syndrome (however, patients with limited allergies such as contact dermatitis or minor allergy to penicillin are acceptable).
5. Any of the following laboratory abnormalities at Visit 1:

   1. Clinically significant ECG abnormality, including prolonged QTc (defined as QTcB > 450 msec),
   2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 1.5 times the upper limit of normal (ULN),
   3. Clinically significant abnormal white blood cell (WBC), absolute neutrophil, or platelet count values,
   4. Any other clinically significant laboratory value.
6. Exposure to an investigational drug within the 30 days prior to Visit 1 or exposure ever to perampanel.
7. Females who are pregnant, lactating, or planning to become pregnant during the study.
8. Use of any medication known to be a strong inducer of CYP3A4 activity within 4 weeks prior to Visit 1; use of CYP3A4 inducers is prohibited for the entire study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Mann, MD, Study Director — Eisai Inc.
Locations (47):
- United States (42):
  - Peoria, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Los Angeles, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Boulder, Colorado
  - Denver, Colorado
  - Milford, Connecticut
  - Boca Raton, Florida
  - Bradenton, Florida
  - Daytona Beach, Florida
  - Delray Beach, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Kissimmee, Florida
  - Largo, Florida
  - Miami, Florida
  - Naples, Florida
  - Orlando, Florida
  - Palm Beach Gardens, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Sunrise, Florida
  - Tampa, Florida
  - Pain and Rehabilitation Clinic of Chicago, Chicago, Illinois
  - Chicago, Illinois
  - Towson, Maryland
  - Boston, Massachusetts
  - West Yarmouth, Massachusetts
  - Southfield, Michigan
  - Missoula, Montana
  - Las Vegas, Nevada
  - Brooklyn, New York
  - High Point, North Carolina
  - Winston-Salem, North Carolina
  - Kettering, Ohio
  - Bensalem, Pennsylvania
  - Norristown, Pennsylvania
  - Warwick, Rhode Island
  - Dallas, Texas
- Canada (5):
  - Kelowna, British Columbia
  - Sarnia, Ontario
  - Toronto, Ontario
  - Pointe-Claire, Quebec
  - Saskatoon, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Cohort 1; Placebo Cohort 2: Placebo (Cohort 1 and 2 differed only in timing of their scheduled visits. Cohort 1 was scheduled to visit every 3 weeks. Cohort 2 was scheduled to visit every week for the first 6 weeks and every 3 weeks thereafter)
- Perampanel Cohort 1, 3-week Titration: Perampanel 8mg (Subjects started at 2mg/day at Baseline and were up-titrated at 3-week intervals by 2mg steps to a total of 8mg or MTD [maximum tolerated dose] and continued at this dose until Week 15)
- Perampanel Cohort 2, 1-week Titration: Perampanel 8mg (Subjects started at 2mg/day at Baseline and were up-titrated at 1-week intervals by 2mg steps to a total of 8mg or MTD and continued at this dose until Week 15)
- Perampanel Cohort 2, 2- Week Titration: Perampanel 8mg (Subjects started at 2mg/day at Baseline and were up-titrated at 2-week intervals by 2mg steps to a total of 8mg or MTD and continued at this dose until Week 15)
Period: Overall Study
Arm/Group | Placebo Cohort 1 | Perampanel Cohort 1, 3-week Titration | Placebo Cohort 2 | Perampanel Cohort 2, 1-week Titration | Perampanel Cohort 2, 2- Week Titration
Started | 26 | 53 | 22 | 22 | 23
Completed | 15 | 21 | 18 | 8 | 9
Not Completed | 11 | 32 | 4 | 14 | 14
Not completed — Adverse Event | 5 | 19 | 2 | 14 | 8
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 7 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 3 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 1
Not completed — Other | 0 | 1 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Cohort 1 | Perampanel Cohort 1, 3-week Titration | Placebo Cohort 2 | Perampanel Cohort 2, 1-week Titration | Perampanel Cohort 2, 2- Week Titration | Total
Number analyzed (Participants) | 26 | 53 | 22 | 22 | 23 | 146
Age, Customized [Number; unit: Participants] — Safety population
  Participants
    <65 years | 10 | 15 | 6 | 2 | 9 | 42
    ≥65 to <75 years | 8 | 15 | 5 | 4 | 3 | 35
    ≥75 years | 8 | 23 | 11 | 16 | 11 | 69
Sex: Female, Male [Count of Participants; unit: Participants] — Safety population-subjects who were randomized, took at least 1 dose of study drug, and had at least 1 post-baseline assessment
  Participants
    Female | 11 | 31 | 8 | 11 | 14 | 75
    Male | 15 | 22 | 14 | 11 | 9 | 71
Race/Ethnicity, Customized [Number; unit: Participants] — Race (Safety population)
  Participants
    White | 25 | 43 | 20 | 21 | 18 | 127
    Black | 1 | 7 | 0 | 0 | 1 | 9
    Asian | 0 | 0 | 0 | 0 | 3 | 3
    Other | 0 | 3 | 2 | 1 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Pain Scores to Week 15/ End of Treatment (EOT) (Including Modified BOCF Data)
Description: Average pain scores are based on pain intensity (11-point Likert-type numerical scale, where 0=no pain and 10=worst possible pain), reported by the subjects in a daily diary. The average pain score for baseline was calculated using the average of the last 7 scores prior to randomization, and the average pain score for Week 15 was computed using the average of the last 7 on-treatment scores prior to Week 15, and they were reported by treatment group.
Time Frame: Baseline and Week 15
Population: Intent-to-Treat (ITT) Population- group of subjects who were randomized, took study drug, and had at least 1 efficacy assessment at Baseline. The modified Baseline Observation Carried Forward (BOCF) method was used.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo Cohort 1 | Perampanel Cohort 1, 3-week Titration | Placebo Cohort 2 | Perampanel Cohort 2, 1-week Titration | Perampanel Cohort 2, 2- Week Titration
Number analyzed (Participants) | 26 | 53 | 22 | 22 | 23
Scores on a scale | -0.55 (1.56) | -1.30 (2.13) | -0.95 (1.77) | -0.50 (1.35) | -1.01 (1.52)

2. Primary Outcome: Responder Rate: Subjects With at Least 30 Percent Reduction in Pain
Description: A responder was a participant with at least 30 percent reduction in average pain scores, using modified BOCF, based on pain intensity (11-point Likert-type numerical scale where 0=no pain and 10=worst possible pain), reported by the subjects in a daily diary. The average pain score for baseline was calculated using the average of the last 7 scores prior to randomization, and the average pain score for Week 15 was computed using the average of the last 7 on-treatment scores prior to Week 15, and they were reported by treatment group.
Time Frame: Baseline and Week 15
Population: ITT Population (Modified BOCF)
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Cohort 1 | Perampanel Cohort 1, 3-week Titration | Placebo Cohort 2 | Perampanel Cohort 2, 1-week Titration | Perampanel Cohort 2, 2- Week Titration
Number analyzed (Participants) | 26 | 53 | 22 | 22 | 23
Percentage of Participants
  Responders (Yes) | 19.2 | 28.3 | 22.7 | 13.6 | 26.1
  Non-Responders (No) | 80.8 | 71.7 | 77.3 | 86.4 | 73.9

3. Primary Outcome: Responder Rate: Subjects With at Least 50 Percent Reduction in Pain
Description: A responder was a participant with at least 50 percent reduction in average pain scores, using modified BOCF, based on pain intensity (11-point Likert-type numerical scale where 0=no pain and 10=worst possible pain), reported by the subjects in a daily diary. The average pain score for baseline was calculated using the average of the last 7 scores prior to randomization, and the average pain score for Week 15 was computed using the average of the last 7 on-treatment scores prior to Week 15, and they were reported by treatment group.
Time Frame: Baseline and Week 15
Population: ITT Population (Modified BOCF)
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo Cohort 1 | Perampanel Cohort 1, 3-week Titration | Placebo Cohort 2 | Perampanel Cohort 2, 1-week Titration | Perampanel Cohort 2, 2- Week Titration
Number analyzed (Participants) | 26 | 53 | 22 | 22 | 23
Percentage of Participants
  Responders (Yes) | 11.5 | 20.8 | 13.6 | 9.1 | 13.0
  Non-Responders (No) | 88.5 | 79.2 | 86.4 | 90.9 | 87.0

4. Primary Outcome: Change From Baseline in Average Pain Scores by Week
Description: Change from baseline in average pain scores by week based on pain intensity (11-point Likert-type numerical scale where 0=no pain and 10=worst possible pain), reported by the subjects in a daily diary. The average pain scores were calculated as the average of available scores in each week, and were reported by treatment group.
Time Frame: Week 1 through Week 16
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo Cohort 1 | Perampanel Cohort 1, 3-week Titration | Placebo Cohort 2 | Perampanel Cohort 2, 1-week Titration | Perampanel Cohort 2, 2- Week Titration
Number analyzed (Participants) | 26 | 53 | 22 | 22 | 23
Scores on a scale
  Week 1 | -0.25 (0.66) | -0.35 (1.03) | -0.43 (0.88) | -0.44 (0.75) | -0.55 (0.71)
  Week 2 | -0.39 (1.11) | -0.60 (1.29) | -0.64 (1.19) | -0.86 (1.19) | -0.74 (1.23)
  Week 3 | -0.68 (1.20) | -1.01 (1.61) | -0.74 (1.31) | -1.22 (1.53) | -1.19 (1.32)
  Week 4 | -0.82 (1.70) | -1.29 (1.88) | -0.89 (1.48) | -1.64 (1.68) | -1.68 (1.49)
  Week 5 | -1.13 (1.93) | -1.46 (1.93) | -0.74 (1.58) | -1.68 (1.93) | -1.23 (1.43)
  Week 6 | -0.81 (1.37) | -1.39 (1.96) | -0.92 (1.66) | -1.53 (2.23) | -1.31 (1.43)
  Week 7 | -0.80 (1.57) | -1.74 (2.12) | -1.21 (1.74) | -1.52 (2.32) | -1.50 (1.67)
  Week 8 | -0.68 (1.43) | -1.92 (2.32) | -1.03 (1.66) | -1.46 (2.21) | -1.68 (2.01)
  Week 9 | -0.53 (1.43) | -1.99 (2.34) | -1.08 (1.79) | -1.24 (1.88) | -1.73 (2.24)
  Week 10 | -0.88 (1.60) | -2.17 (2.30) | -1.14 (1.92) | -1.48 (1.71) | -1.36 (2.38)
  Week 11 | -0.96 (1.67) | -2.33 (2.28) | -1.01 (1.64) | -1.98 (1.63) | -1.46 (2.51)
  Week 12 | -0.99 (1.78) | -2.52 (2.36) | -1.01 (1.67) | -1.82 (1.43) | -1.40 (2.55)
  Week 13 | -0.80 (1.72) | -2.13 (2.31) | -1.05 (1.78) | -1.77 (1.88) | -1.96 (1.92)
  Week 14 | -1.00 (1.85) | -2.38 (2.27) | -1.17 (1.83) | -1.46 (1.72) | -2.19 (1.91)
  Week 15 | -0.88 (1.96) | -2.42 (2.40) | -1.17 (1.91) | -1.32 (2.00) | -2.09 (1.77)
  Week 16 | -1.79 (1.11) | -3.17 (2.18) | -0.65 (1.93) | -0.88 (1.97) | -0.95 (1.39)

5. Secondary Outcome: Change From Baseline to Week 15/EOT in Average Sleep Interference Scores
Description: The average of the last 7 available sleep scores prior to the visit, based on the 11-point Likert-type numerical rating scale for sleep interference (where 0=pain did not interfere with sleep, to 10=pain completely interfered with sleep [unable to sleep]), and they were reported by treatment group.
Time Frame: Baseline and Week 15
Population: ITT Population (Modified BOCF)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo Cohort 1 | Perampanel Cohort 1, 3-week Titration | Placebo Cohort 2 | Perampanel Cohort 2, 1-week Titration | Perampanel Cohort 2, 2- Week Titration
Number analyzed (Participants) | 26 | 53 | 22 | 22 | 23
Scores on a scale | -0.58 (1.30) | -0.46 (1.92) | -1.16 (1.60) | -0.48 (1.29) | -0.75 (1.41)

6. Secondary Outcome: Patient Global Impression of Change (PGIC) at Week 15/EOT
Description: Changes were calculated using the modified BOCF method
Time Frame: Week 15
Population: Subset of ITT population used, including subjects that completed PGIC at Week 15 visit, and using BOCF (baseline observation carried forward) subjects that terminated prior to Week 15 received a 'No Change' if due to AE or Lack of Therapeutic Efficacy, subjects who discontinued due to other reasons used PGIC scores from Early Termination visit.
Measure: Number; unit: Participants
Arm/Group | Placebo Cohort 1 | Perampanel Cohort 1, 3-week Titration | Placebo Cohort 2 | Perampanel Cohort 2, 1-week Titration | Perampanel Cohort 2, 2- Week Titration
Number analyzed (Participants) | 20 | 42 | 20 | 19 | 22
Participants
  Very much improved | 0 | 4 | 1 | 1 | 1
  Much improved | 3 | 8 | 4 | 2 | 1
  Minimally improved | 1 | 2 | 3 | 2 | 4
  No change | 13 | 27 | 11 | 13 | 15
  Minimally worse | 2 | 0 | 1 | 0 | 1
  Much worse | 1 | 1 | 0 | 1 | 0
  Very much worse | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Clinician Global Impression of Change (CGIC) at Week 15/EOT
Description: Changes were calculated using the modified BOCF method
Time Frame: Week 15
Population: Subset of ITT population used, including subjects that completed CGIC at Week 15 visit, and using BOCF (baseline observation carried forward) subjects that terminated prior to Week 15 received a 'No Change' if due to AE or Lack of Therapeutic Efficacy, subjects who discontinued due to other reasons used CGIC scores from Early Termination visit.
Measure: Number; unit: Participants
Arm/Group | Placebo Cohort 1 | Perampanel Cohort 1, 3-week Titration | Placebo Cohort 2 | Perampanel Cohort 2, 1-week Titration | Perampanel Cohort 2, 2- Week Titration
Number analyzed (Participants) | 21 | 45 | 20 | 21 | 22
Participants
  Very much improved | 1 | 3 | 2 | 0 | 2
  Much improved | 1 | 8 | 2 | 2 | 2
  Minimally improved | 2 | 6 | 2 | 3 | 3
  No change | 16 | 28 | 14 | 16 | 15
  Minimally worse | 1 | 0 | 0 | 0 | 0
  Much worse | 0 | 0 | 0 | 0 | 0
  Very much worse | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline to Week 15/EOT in HADS Anxiety Subscale Scores (Modified BOCF)
Description: The HADS (Hospital Anxiety and Depression Scale) is a widely used, self-reported, 14-item instrument that measures the presence and severity of anxiety and depression. It consists of 2 subscales; a 7-item anxiety subscale (HADS-A) and a 7-item depression subscale (HADS-D). HADS-A consists of a 7-item scale, each scored on a 4-pt scale (0, 1, 2, or 3), where a higher score indicates worse anxiety. Range of possible HADS anxiety subscale scores is 0 to 21, and normal=(0-7), mild=(8-10), moderate=(11-14), and severe=(15-21).
Time Frame: Baseline and Week 15
Population: ITT population (Modified BOCF)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo Cohort 1 | Perampanel Cohort 1, 3-week Titration | Placebo Cohort 2 | Perampanel Cohort 2, 1-week Titration | Perampanel Cohort 2, 2- Week Titration
Number analyzed (Participants) | 26 | 53 | 22 | 22 | 23
Scores on a scale | -0.2 (1.31) | 0.0 (3.25) | 0.1 (2.90) | 0.0 (1.28) | -0.1 (2.35)

9. Secondary Outcome: Change From Baseline to Week 15/EOT in HADS Depression Subscale Scores (Modified BOCF)
Description: The HADS (Hospital Anxiety and Depression Scale) is a widely used, self-reported, 14-item instrument that measures the presence and severity of anxiety and depression. It consists of 2 subscales; a 7-item anxiety subscale (HADS-A) and a 7-item depression subscale (HADS-D). HADS-D consists of a 7-item scale, each scored on a 4-pt scale (0, 1, 2, or 3), where a higher score indicates worse depression. Range of possible HADS depression subscale scores is 0 to 21, and normal=(0-7), mild=(8-10), moderate=(11-14), and severe=(15-21).
Time Frame: Baseline and Week 15
Population: ITT population (Modified BOCF)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo Cohort 1 | Perampanel Cohort 1, 3-week Titration | Placebo Cohort 2 | Perampanel Cohort 2, 1-week Titration | Perampanel Cohort 2, 2- Week Titration
Number analyzed (Participants) | 26 | 53 | 22 | 22 | 23
Scores on a scale | -0.1 (1.51) | 0.1 (2.11) | -0.6 (2.28) | 0.2 (2.66) | -0.3 (1.49)

10. Secondary Outcome: Analysis of Allodynia (Present/Not Present) at Week 15/EOT- by Treatment Groups ITT Population (Modified BOCF)
Description: Allodynia is defined as a painful reaction to a non-painful stimulus.
Time Frame: Week 15
Population: ITT population (Modified BOCF)
Measure: Number; unit: Participants
Arm/Group | Placebo Cohort 1 | Perampanel Cohort 1, 3-week Titration | Placebo Cohort 2 | Perampanel Cohort 2, 1-week Titration | Perampanel Cohort 2, 2- Week Titration
Number analyzed (Participants) | 26 | 53 | 22 | 22 | 23
Participants
  Yes | 22 | 47 | 17 | 17 | 19
  No | 4 | 6 | 5 | 5 | 4

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the time the patient signed the informed consent form until 30 days after the last dose of study drug.
Description: Safety variables included AEs, laboratory values, vital signs, and electrocardiogram measurements.
Arm/Group | Placebo Cohort 1 | Perampanel Cohort 1, 3-week Titration | Placebo Cohort 2 | Perampanel Cohort 2, 1-week Titration | Perampanel Cohort 2, 2- Week Titration
Serious Adverse Events (participants affected / at risk) | 1/26 | 7/53 | 2/22 | 1/22 | 1/23
Other Adverse Events (participants affected / at risk) | 11/26 | 36/53 | 14/22 | 18/22 | 16/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Cohort 1 (N=26) | Perampanel Cohort 1, 3-week Titration (N=53) | Placebo Cohort 2 (N=22) | Perampanel Cohort 2, 1-week Titration (N=22) | Perampanel Cohort 2, 2- Week Titration (N=23)
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Vestibulitis (General disorders) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Carotid artery occlusion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Cohort 1 (N=26) | Perampanel Cohort 1, 3-week Titration (N=53) | Placebo Cohort 2 (N=22) | Perampanel Cohort 2, 1-week Titration (N=22) | Perampanel Cohort 2, 2- Week Titration (N=23)
Vision blurred (Eye disorders) | 0 | 0 | 0 | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 3 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 3 | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 1 | 3 | 2
Gait disturbance (General disorders) | 0 | 2 | 0 | 7 | 2
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 2 | 0 | 2 | 2
Dizziness (Nervous system disorders) | 8 | 22 | 1 | 12 | 8
Dysarthria (Nervous system disorders) | 0 | 2 | 0 | 4 | 1
Headache (Nervous system disorders) | 2 | 4 | 1 | 3 | 1
Somnolence (Nervous system disorders) | 1 | 9 | 4 | 2 | 5
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 3 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 1 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No